CLINICAL TRIAL: NCT01354483
Title: Feasibility and Safety of Umbilical Cord Blood Cell Transplant Into Injured Spinal Cord: an Open-Labeled, Dose-Escalating Clinical Trial
Brief Title: Umbilical Cord Blood Mononuclear Cell Transplant to Treat Chronic Spinal Cord Injury
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: China Spinal Cord Injury Network (Network)
Collaborators: Chengdu PLA General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: CN102B_KM
Record Dates: First submitted 2011-02-14; First posted 2011-05-17 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injury; umbilical cord blood mononuclear cell; lithium carbonate
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Methylprednisolone; Lithium Carbonate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- Treatment Group A (Experimental): Umbilical cord blood mononuclear cell, 1.6 million
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Treatment Group B (Experimental): Umbilical cord blood mononuclear cell, 3.2 million
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Treatment Group C (Experimental): Umbilical cord blood mononuclear cell, 6.4 million
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell
- Treatment Group D (Experimental): Umbilical cord blood mononuclear cell, 6.4 million; mehtylprednisolone
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell; Biological: Methylprednisolone
- Treatment Group E (Experimental): Umbilical cord blood mononuclear cell, 6.4 million; methylprednisolone; 6 week course of lithium carbonate tablet
  Interventions: Biological: Umbilical Cord Blood Mononuclear Cell; Biological: Methylprednisolone; Drug: Lithium Carbonate Tablet

INTERVENTIONS:
Biological: Umbilical Cord Blood Mononuclear Cell
Biological: Methylprednisolone — 30mg/kg i.v. methylprednisolone
  Arms: Treatment Group D; Treatment Group E
Drug: Lithium Carbonate Tablet — 6 weeks
  Arms: Treatment Group E

SUMMARY:
The purpose of this study is to investigate the feasibility, safety, efficacy and optimal dose of umbilical cord blood mononuclear cell transplant in the treatment of chronic spinal cord injuries.

DETAILED DESCRIPTION:
This is an open-label dose-escalating clinical trial. 20 patients will be randomly divided into 5 groups, 4 patient per group. The first three groups of four patients will receive transplants of increasing dose of HLA-matched umbilical cord blood mononuclear cells, starting from 4 spinal cord injection of 4µL of cell suspensions in Group A to 8µL in Group B and 16µL in Group C. If more than one subjects show neurological loss attributable to the cell injections, the trial will fall back to the previous dose. In the Group D, the highest volume of cells that do not cause neurological deficits (e.g. 16µL x4) along with a single bolus of 30 mg/kg methylprednisolone sodium succinate (MPSS) will be provided. Subjects in the Group E receive the same treatment as Group D plus a 6-week course of oral lithium carbonate. All subjects will enroll for three months intensive rehabilitation after the cell transplant.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with chronic spinal cord injury (>12 months post-initial spinal cord injury surgery) with stable neurologic findings for at least 6 months
* Subjects with current neurological status of ASIA A
* The neurological level of the subjects is between C5 and T11
* The injured site of the spinal cord is within three vertebral levels
* Subjects must be able to read, understand, and complete the VAS
* Subjects who have voluntarily signed and dated an informed consent form prior to any study procedures.

Exclusion Criteria:

* Significant renal, cardiovascular, hepatic and psychiatric diseases
* Significant medical diseases or infection
* Pregnant or lactating woman
* Female of childbearing potential and who is unwilling to use an effective contraceptive method while enrolled in the study
* The length of spinal cord lesion exceeds three segments
* Unavailability of HLA matched umbilical cord blood cells
* any contraindication of laminectomy operation, methylprednisolone and/or lithium carbonate
* Subject who is currently participating in another investigational study or has been taking any investigation drug within the last 4 weeks prior to screening of the study
* In opinion of the investigator, who suggests that the subject would not be compliant with the study protocol and/or would not be suitable to participate the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2013-09 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes from Baseline in ASIA motor and sensory scores | Day 0, 3, Week 1, 2, 6, 14, 24, 48

SECONDARY OUTCOMES:
Spinal Cord Independence Measure (SCIM) score | Week 0, 2, 6, 14, 24, 48
Walking Index of Spinal Cord Injury (WISCI) Level | Week 0, 2, 6, 14, 24 and 48
Kunming Walking Score | Week 0, 2, 6, 14, 24, 48
Modified Ashworth Scale (MAS)of spasticity | Day 0, 3, Week 1, 2, 6, 14, 24 48
Visual Analog Scale of pain | Day 0, 3, Week 1, 2, 6, 14, 24, 48

CONTACTS AND LOCATIONS:
Overall Officials: Hui Zhu, MD, Principal Investigator — Chengdu PLA General Hospital
Locations (1):
- Treating Center of Spinal Cord Injury, Chengdu Army Kunming General Hospital, Kunming, Yunnan, China